CLINICAL TRIAL: NCT05125874
Title: A Clinical Study to Evaluate the Immunogenicity and Safety of Sequential Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Against COVID-19 in Healthy Adults Aged 18 Years and Older After the Vaccination of 2 Doses of Inactivated Vaccines
Brief Title: Clinical Study for Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Booster Immunization
Acronym: COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICV-V-01-Booster
Record Dates: First submitted 2021-11-09; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Pandemic
Keywords: V-01 Booster
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-01 COVID-19 Vaccine (Experimental): One dose administrated by intramuscular injection
  Interventions: Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Fusion Protein Vaccine — The product should be a milky-white suspension for injection. For prevention of SARS-CoV-2 infection.
  Other Names: V-01

SUMMARY:
A Clinical Study to Evaluate the Immunogenicity and Safety of Sequential Immunization of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Against COVID-19 in Healthy Adults Aged 18 Years and Older After the Vaccination of 2 Doses of Inactivated Vaccines

DETAILED DESCRIPTION:
This is a single arm, open-label clinical study. 45 participants aged 18 years and older who have completed the 2 doses of administration of inactive vaccines will be enrolled in this study to evaluate the safety and immunogenicity of V-01.

The participants will be collected blood before immunization, on day 7, day 14, day 28 and 6 month to evaluate humoral immunity.

All adverse events (AEs) within 30 minutes and 0-7 days after booster immunization, and unsolicited AEs from 8 to 28 days after booster immunization, as well as SAEs and AESIs from the first vaccination to 12 months after booster immunization will be collected from all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years and older who have completed the second dose of 2-dose regimen of inactive vaccination (Vero cell) against SARS-CoV-2 in the past 3-6 months;
2. Voluntarily participate in the study and sign the informed consent form, who can provide valid ID and follow the study protocol requirement;
3. In the past 14 days, no history of high or medium risk of the epidemic, overseas travel history or residence history; no history of contact with confirmed, asymptomatic or suspected COVID-19 cases; no history of contact with the persons from high- and medium-risk epidemic areas or contact patients with fever or respiratory symptoms; and those who are not in isolation period.
4. Males of reproductive potential and females of childbearing potential voluntarily agree to take effective and acceptable contraceptive methods from the signing of informed consent form to 3 months after vaccination.

Exclusion Criteria:

1. Confirmed COVID-19 cases, or positive for SARS-CoV-2 test by RT-PCR.
2. History of previous COVID-19 infection.
3. Fever is suspected or diagnosed within 72 hours before enrollment, or the axillary body temperature ≥37.3℃ on the day of enrollment.
4. History of severe allergy to any vaccine, e.g., acute allergic reactions, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain etc., or be allergic to any components of V-01.
5. People who currently suffer from the following diseases:

   1. Symptoms related to acute respiratory infections (such as: sneezing, nasal congestion, runny nose, cough, sore throat, loss of taste, chills, shortness of breath, etc.)
   2. Patients with thrombocytopenia, any coagulation dysfunction, or receive anticoagulant treatment, etc.
   3. Patients with congenital or acquired angioedema/neuroedema;
   4. A history of congenital or acquired immunodeficiency or autoimmune disease (except for mild psoriasis, controllable autoimmune thyroid disease, vitiligo, or stable celiac disease that does not require immunosuppressive or immunomodulatory therapy); no spleen , or history of spleen surgery, history of trauma, or treatment with immunomodulators within 6 months, such as: glucocorticoid with the dose causing immunosuppressive (dose reference: equivalent to prednisone 20mg/day, more than one week); or monoclonal antibody ; or thymosin; or interferon, etc.; but local medication (such as ointment, eye drops, inhalation or nasal spray) is allowed.
   5. Patients with active tuberculosis, viral hepatitis, human immunodeficiency virus or syphilis infection.
   6. Patients with acute diseases, or acute attacks of chronic diseases, or uncontrolled severe chronic diseases: history of chronic respiratory diseases (including moderate to severe asthma, COPD, pulmonary fibrosis), hypertension that cannot be controlled by drugs (systolic blood pressure ≥150mmHg) And/or diastolic blood pressure ≥100mmHg), history of severe cardiovascular disease (including heart failure, coronary artery disease, cardiomyopathy), history of chronic kidney disease, history of cancer (except for basal cell carcinoma), diabetes (unsatisfied blood sugar control or diabetes related serious complications).
6. Received attenuated live vaccine within 28 days before the vaccination or any subunit vaccines and inactivated vaccines within 14 days before the vaccination.
7. Injection of immunoglobulin and/or other blood products within 3 months before the administration of study vaccine; or with the plan to use such product within 6 month after immunization.
8. Pregnant (including positive urine pregnancy test for women of childbearing age) or breastfeeding women. Or women or their partners who have a pregnancy plan within 3 months after the trial vaccination.
9. Have participated in or are participating in other COVID-19 related clinical trials, or are participating in other drug clinical trials;
10. Those considered by the investigator as inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Seroconvension of SARS-CoV-2 neutralizing antibodies | 14 days and 28 days after booster immunization
  The seroconvension of SARS-CoV-2 neutralizing antibodies on 14 days and 28 days after booster immunization
GMT of SARS-CoV-2 neutralizing antibodies | 14 days and 28 days after booster immunization
  The GMT of SARS-CoV-2 neutralizing antibodies on 14 days and 28 days after booster immunization
GMI of SARS-CoV-2 neutralizing antibodies | 14 days and 28 days after booster immunization
  The GMI of SARS-CoV-2 neutralizing antibodies on 14 days and 28 days after booster immunization

SECONDARY OUTCOMES:
GMT of SARS-CoV-2 (wild type) neutralizing antibodies | Before and on day 7 after booster immunization
  GMT of SARS-CoV-2 (wild type) neutralizing antibodies before and on day 7 after booster immunization
Seroconvension of SARS-CoV-2 (wild type) neutralizing antibodies | On day 7 after booster immunization
  The seroconvension of SARS-CoV-2 (wild type) neutralizing antibodies on day 7 after booster immunization
GMI of SARS-CoV-2 (wild type) neutralizing antibodies | On day 7 after booster immunization
  The GMI of SARS-CoV-2 (wild type) neutralizing antibodies on day 7 after booster immunization
GMT of SARS-CoV-2 delta variant (B1.617.2) neutralizing antibodies | Before and on day 7, day 14, day 28 after booster immunization
  The GMT of SARS-CoV-2 delta variant (B1.617.2) neutralizing antibodies before and on day 7, day 14, day 28 after booster immunization
Seroconvension of SARS-CoV-2 delta variant (B1.617.2) neutralizing antibodies | On day 7, day 14, day 28 after booster immunization
  The seroconvension of SARS-CoV-2 delta variant (B1.617.2) neutralizing antibodies on day 7, day 14, day 28 after booster immunization
GMI of SARS-CoV-2 delta variant (B1.617.2) neutralizing antibodies | On day 7, day 14, day 28 after booster immunization
  The GMI of SARS-CoV-2 delta variant (B1.617.2) neutralizing antibodies on day 7, day 14, day 28 after booster immunization
Long-term immunity | 6 months after booster immunization
  The seroconvension, GMT and GMI of SARS-CoV-2 (wild type) and SARS-CoV-2 delta variant (B1.617.2) neutralizing antibodies after 6 months after booster immunization
Incidence of AEs | 30 minutes, 0-7 days, 8-28 days after booster immunization, 12 months after booster immunization.
  The incidence of adverse events (AEs) occur within 30 minutes, 0-7 days, 8-28 days after booster immunization, as well as SAEs and AESIs from the first vaccination to 12 months after booster immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Ligong Lu, Dr., Principal Investigator — Zhuhai People's Hospital Medical Group
Locations (1):
- Zhuhai Peoples' Hospital Medical Group, Zhuhai, Guangdong, China